CLINICAL TRIAL: NCT06492837
Title: A Phase II Trial Investigating MOsunetuzumab and ZAnubrutinib (BGB-3111) in Relapsed/refracTory Follicular Lymphoma Patients (MOZART)
Brief Title: Study With Mosunetuzumab and Zanubrutinib in R/R Follicular Lymphoma Patients
Acronym: FIL_MOZART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_MOZART
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; Mosunetuzumab; Zanubrutinib; Relapsed/refractory follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mosunetuzumab in combination with Zanubrutinib (Experimental): Pre-phase: Zanubrutinib 320 mg daily by mouth (D-15 to D-1)
  Induction phase cycle 1 (Q21 days):
  * Zanubrutinib 320 mg daily by mouth (D1-21)
  * Mosunetuzumab 5 mg, SC (D1)
  * Mosunetuzumab 45 mg, SC (D8)
  * Mosunetuzumab 45 mg, SC (D15)
  Induction phase cycles 2-12 (Q28 days):
  * Zanubrutinib 320 mg daily by mouth (D1-28)
  * Mosunetuzumab 45 mg, SC (D1)
  Maintenance phase cycles 13-24 (Q28 days): Zanubrutinib 320 mg daily by mouth (D1-28)
  Tocilizumab will be administered as needed to manage cytokine release syndrome (CRS) events.
  Interventions: Drug: Mosunetuzumab in combination with Zanubrutinib

INTERVENTIONS:
Drug: Mosunetuzumab in combination with Zanubrutinib — Combinations of Mosunetuzumab and Zanubrutinib as salvage strategy in patients with relapsed/refractory follicular lymphoma who have received at least one line of prior systemic therapy.
  Other Names: LUNSUMIO in combination with BRUSINKA

SUMMARY:
This is a Phase 2, multicenter study evaluating the efficacy and safety of mosunetuzumab + zanubrutinib (M+Z) used as salvage strategy in patients with R/R FL who have received at least one line of prior systemic therapy.

DETAILED DESCRIPTION:
Eligible patients receive a pre-phase with oral zanubrutinib followed by an induction phase with mosunetuzumab combined with oral zanubrutinib.

Patients responsive to induction phase with M+Z (C1-12) and achieving at least SD will receive maintenance with zanubrutinib for additional 12 months (C13-24).

There will be an initial safety run-in (SRI) phase of 10 patients which will be closely monitored for the observed toxicities during the first three cycles of induction (from C1D1 to C3D28). No patients will be further enrolled until SRI analyses is completed.

If no unexpected toxicity has been observed, subsequent patients will be monitored only for patient informed consent, grade 3-5 toxicities and SAEs as well as remission status.

Safety data will be evaluated by an independent data safety monitoring board (DSMB) that will advise the principal investigators on the continuation of the study. Safety events will be analyzed and compared with the previously described safety profile of mosunetuzumab alone and other bispecific-containing regimens to exclude the risk of potential toxicity for all study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent form approved by the National Ethics Committee (NEC) prior to the initiation of any screening or study-specific procedures and able to understand and to comply with the requirements of the study and the schedule of assessments.
2. Histologically documented diagnosis of cFL (CD20+ by flow cytometry or immunohistochemistry) as defined in the International Consensus Classification of Mature Lymphoid Neoplasms (Campo E., 2022) and in the World Health Organization Classification (WHO) 5th edition 2022.
3. Age ≥18 years.
4. Relapsed or refractory disease. Histologic confirmation of FL relapse is not mandatory but is highly recommended.
5. At least one and up to three lines of systemic therapy containing an anti-CD20 antibody (anti-CD20 alone and/or in combination with radiotherapy is not considered as a line of therapy).
6. FL requiring systemic therapy assessed by investigator based on tumor size and/or Groupe d'Etude des Lymphomes Folliculaires criteria.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
8. Availability of histological material for centralized revision. Central pathology review is not mandatory for start of treatment.
9. At least one measurable or evaluable site of disease at relapse as documented by CT scan (nodes ≥ 1.5 cm in the longest transverse diameter) or FDG-PET (avid FDG sites). Note: MRI is allowed only if CT scan cannot be performed. Patients with exclusive bone marrow involvement are eligible.
10. Adequate hematological counts defined as follows:

    * Absolute neutrophil count (ANC) > 1.0 x 109/L;
    * Platelet count ≥ 75 x 109/L;
    * Hemoglobin ≥ 9 g/dL.
11. Adequate renal function defined as creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula, normalized to 1.72 m2).
12. Adequate hepatic function per local laboratory reference range as follows:

    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN;
    * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin).
13. Subject must be able to adhere to the study visit schedule and other protocol requirements.
14. Subject must be able to swallow capsules or tablets.
15. Women must be:

    * postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months);
    * surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy);
    * if they are childbearing potential, completely abstinent (periodic abstinence is not permitted) or if sexually active, be practicing a highly effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double barrier method (e.g.: condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization), before entry, and must agree to continue to use the same method of contraception throughout the study and for 30 days after receiving the last dose of zanubrutinib and 3 months after receiving the last dose of mosunetuzumab.
16. Women of childbearing potential must have a negative pregnancy test at screening.
17. Men must agree to use an acceptable method of contraception for the duration of the study and for 1 week after receiving the last dose of study drug.
18. Male even if surgically sterilized (i.e., status post vasectomy) must agree to 1 of the following:

    * practice effective barrier contraception (e.g.: condoms) , or
    * agree to practice abstinence, when this is in line with the usual lifestyle of the subject (periodic abstinence is not permitted).

Exclusion Criteria:

1. Histological diagnosis different from cFL (Campo E., 2022).
2. R/R FL who were treated with more than three lines of previous treatment (autologous stem cell transplant performed as part of consolidation to a previous line of therapy should not be considered as a line of therapy; rituximab maintenance as part of a previous line of therapy should not be considered as a line of therapy; radiotherapy alone or in combination with rituximab is not considered a line of therapy).
3. Patients with stage I or II (limited stage) suitable for RT alone treatment.
4. Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor (BTKi).
5. Prior exposure to an anti-CD20xCD3 bispecific antibody (bsAbs).
6. Need of anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon). Requires ongoing treatment with a strong CYP3A inducer.
7. Evidence or any history of transformation from FL to other aggressive histology.
8. Prior allogeneic hematopoietic stem cell transplantation.
9. History of severe bleeding disorder (G>3), or history of spontaneous bleeding requiring blood transfusion or other medical intervention. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug
10. Life expectancy < 6 months.
11. History of progressive multifocal leukoencephalopathy (PML).
12. History of hemophagocytic lymphohistiocytosis (HLH) or chronic active EBV.
13. History of autoimmune disease, including, but not limited to: myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
14. Primary central nervous system (CNS) lymphoma or CNS involvement by lymphoma at screening as confirmed by mandatory brain computed tomography (CT) scan and, if clinically indicated, by lumbar puncture.
15. Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, investigational therapy, including targeted small molecule agents within 14 days prior to the first dose of study drug. If receiving glucocorticoid treatment at screening, must be a maximum daily dose of prednisone 10 mg (or equivalent).
16. Prior treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 90 days prior to first therapy administration.
17. Any uncontrolled or significant cardiovascular disease [NYHA class ≥2].

    1. Myocardial infarction within 6 months before screening
    2. Unstable angina within 3 months before screening
    3. New York Heart Association class III or IV congestive heart failure
    4. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes)
18. Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent.
19. Any history of other active malignancies within 3 years prior to study entry, except for adequately treated in situ carcinoma of the uterine cervix, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, non-muscle-invasive bladder cancer, localized Gleason score 6 prostate cancer, previous malignancy confined and surgically resected with curative intent.
20. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

    1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal), including active ongoing infection from SARS-CoV-2;
    2. Chronic or acute hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen (Ag) negative, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from previous infection or intravenous immunoglobulins (IVIG) may participate; inactive carriers (HBsAg positive with undetectable HBV- DNA) are eligible. Patients with presence of HCV antibody are eligible only if PCR negative for HCV-RNA;
21. HIV seropositivity.
22. Pregnant or lactating women. If female, the patient is pregnant or breast-feeding.
23. Severe or debilitating pulmonary disease.
24. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
25. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs.
26. Major surgery within 4 weeks of the first dose of study drug.
27. Vaccination or requirement for vaccination with a live vaccine within 28 days prior to the first dose of study drug or at any time during planned study treatment.
28. Ongoing alcohol or drug addiction or any psychiatric condition(s) which would compromise ability to comply with study procedures.
29. Hypersensitivity to zanubrutinib or mosunetuzumab or any of the other ingredients of the applicable study drugs.
30. Active and/or ongoing autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2033-09-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | 36 months
  CRR at the end of the induction therapy

SECONDARY OUTCOMES:
Overall Response Rate (ORR), Partial Response (PR) Rate at the end of induction treatment (EOI) | 36 months
  ORR and PR Rate at the end of induction treatment (EOI)
Overall Response Rate (ORR), Partial Response (PR) Rate at the end of maintenance (EOT, end of treatment) | 48 months
  ORR and PR Rate at the end of maintenance (EOT, end of treatment)
Progression Free Survival (PFS) | 108 months
  PFS defined as the time between the start of prephase and the first documentation of recurrence, progression or death from any cause.
Overall Survival (OS) | 108 months
  OS defined as the time between the start of prephase and death from any cause.
Duration of Response (DOR) | 108 months
  DOR defined as the time from the first documentation of tumor response (CR or PR) to disease progression or death from any cause
Duration of Complete Response (DOCR) | 108 months
  DOCR defined as the time from the first documentation of tumor complete response to disease progression or death from any cause.
Time-to-next-treatment (TTNT) | 108 months
  TTNT defined as the time between start of prephase and the initiation of the next line of therapy.
Event free survival (EFS) | 108 months
  EFS defined as the time from the start of prephase to disease progression, death, or discontinuation of treatment for any reason (e.g. toxicity, patient preference), or initiation of a new treatment without documented progression.
Frequency and severity of Adverse Events (AEs) and Serious AEs (SAEs) | 108 months
  AEs and SAEs classified as per the latest version of CTCAE.
Frequency and severity of cytokine release syndrome (CRS) and Neurological Adverse Events (NAE) | 36 months
  CRS and NAE will be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) Grading Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ladetto, Prof, Principal Investigator — Department of Translational Medicine of the Università degli Studi del Piemonte Orientale, Novara, Italy. AO SS Antonio e Biagio e C. Arrigo, Alessandria, Italy.; Stefano Luminari, Prof, Principal Investigator — Oncology and Regenerative Medicine, University of Modena and Reggio Emilia, Modena, Italy. Hematology Unit of AUSL-IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Emilia, Italy.
Locations (24):
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Liverpool Hospital, Liverpool
  - St. Vincent Hospital Melbourne, Melbourne
  - Princess Alexandra Hospital, Woolloongabba
- Italy (20):
  - Fondazione del Piemonte per l'Oncologia - IRCCS, Ematologia, Candiolo, Torino
  - AOU SS. Antonio e Biagio e Cesare Arrigo, SCDU Ematologia, Alessandria
  - AOU Ospedali Riuniti, Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S.Giuseppe Moscati, S.C. Ematologia e Trapianto emopoietico, Avellino
  - IRCCS Istituto Tumori Giovanni Paolo II, U.O.C Ematologia, Bari
  - Policlinico S.Orsola-Malpighi, Istituto di Ematologia "Seragnoli", Bologna
  - ASST Spedali Civili di Brescia, Ematologia, Brescia
  - Azienda Ospedaliera Universitaria Policlinico - S. Marco, UOC di Ematologia, Catania
  - Azienda Ospedaliera Universitaria Careggi, Unità funzionale di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda, SC Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Ematologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Ematologia, Monza
  - AOU Maggiore della Carità di Novara, SCDU Ematologia, Novara
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Divisione di Ematologia, Palermo
  - Azienda USL Piacenza, UOC Ematologia e Centro Trapianti, Piacenza
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Ematologia, Reggio Emilia
  - Ospedale degli Infermi di Rimini, U.O. di Ematologia, Rimini
  - Policlinico Umberto I - Università La Sapienza, Istituto Ematologia, Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, S.C.Ematologia, Torino
  - Ospedale Ca' Foncello, S.C di Ematologia, Treviso

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may contact the FIL board at segreteriadirezione@filinf.it to share invidual-level patients' clinical data analysed for this manuscript (for the avoidance of doubt, no identifiable data, such as name, address, hospital name, date of birth, or any other identifying data, will be shared and should not be requested).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In compliance with the domestic ethics guideline and applicable legislation, invidual deindentified patients' data underlying the results reported in the publication article (including study protocol, statistical analysis plan and data coding) can be shared until 5 years after the publication of the article.
Access Criteria: For each data sharing request, it is essential that a proforma (available on request) is completed that describes the general purpose, specific aims, data items requested, analysis plan and acknowledgment of the trial management team. Requests will be reviewed based on scientific merit and ethical principles. Requestors who are granted access to the data will be required to complete a data sharing agreement that will be signed by the requester and FIL.